CLINICAL TRIAL: NCT01191749
Title: Phase II Pilot Study Of Alemtuzumab In Patients With Low Or INT-1 Risk Myelodysplastic Syndrome (MDS), Aplastic Anemia (AA), Or T-Cell Large Granular Lymphocytic Leukemia (T-LGL)
Brief Title: Alemtuzumab in Myelodysplastic Syndrome (MDS), Aplastic Anemia, and T-Cell Large Granular Lymphocytic Leukemia (T-GL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0187
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Leukemia
Keywords: Hematologic Disorder; Aplastic Anemia; T - Cell Large Granular Lymphocytic Leukemia; T-LGL; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; CLL; Chemotherapy; Alemtuzumab
MeSH Terms: conditions — Leukemia; Hematologic Diseases; Anemia, Aplastic; Leukemia, Large Granular Lymphocytic; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alemtuzumab (Experimental): Alemtuzumab 10 mg by vein over 2 hours on Days 1 to 10 of a 28 day cycle.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — 10 mg by vein over 2 hours on Days 1 to 10 of a 28 day cycle.
  Other Names: CAMPATH-1H; Campath

SUMMARY:
The goal of this clinical research study is to determine the effectiveness of alemtuzumab in patients with aplastic anemia, MDS, or T-Cell large granular lymphocytic leukemia. The safety of alemtuzumab will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Alemtuzumab is designed to attach to a protein that is found on certain immune cells, which may cause the cell to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive alemtuzumab on Days 1-10 of one 28-day cycle. It will be given either by vein over 2 hours or by injection under the skin 1 time a day. Your doctor will tell you how the drug will be given.

In order to get alemtuzumab provided for your treatment, the study staff will be filling out a form with your name and medical information (protected health information) for the company as part of the Campath Distribution Program.

All participants will receive the same dose of alemtuzumab unless the starting dose causes intolerable side effects. If this happens, all future participants will receive a lower dose.

Depending on your doctor's decision, to lower the risk of side effects you will receive Tylenol (acetaminophen) and Benadryl (diphenhydramine) or other drugs such as steroids (either by mouth or by a short infusion by vein), 30 minutes before each alemtuzumab dose.

If you are receiving alemtuzumab and have chills during the infusion, you may receive Demerol (meperidine hydrochloride, a painkiller) to help control them.

Starting on Day 1 and continuing at least 8 weeks after the last dose of study drug, you will be given 2 antibiotics to help fight infection. You will take Valacyclovir (or a similar drug) 1 time each day. You will take Trimethoprim/Sulfamethoxazole (or a similar drug) 2 times a day, 3 times per week. You will take both antibiotics by mouth.

Study Visits:

At Week 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.

At Weeks 2-4, blood (about 1 tablespoon) will be drawn for routine tests.

Beginning at Week 5 (+/- 3 days) and then 1 time monthly:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.

At Week 12 (+/- 3 days) (end of the 3rd month), you will have a bone marrow aspiration and/or biopsy to test for chromosome abnormalities (if chromosomes were abnormal at screening) and to check the status of the disease. You may have additional bone marrow aspirations or biopsies if your doctor feels they are necessary.

You will be asked about any side effects you may be having at each of your study visits. At any time during the study, if the doctor thinks it is needed, you will have a chest x-ray, a CT scan, or a PET scan to check the status of the disease.

Length of Study:

You will receive only one cycle of the study drug. Your participation on the study will be over after you have completed the end-of-study visit. You will be taken off study early if the disease gets worse or intolerable side effects occur.

End-of Study-Visit:

When you come off study you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will have a bone marrow aspiration and/or biopsy to check for chromosome abnormalities, test for low levels of leukemia or lymphoma, to check the status of the disease, and molecular testing. Molecular tests are designed to look at the way the different parts of a cell (including DNA, RNA, and proteins) work together.
* Blood (about 2 teaspoons) will be drawn to check levels of T-cells and immunoglobulins.

This is an investigational study. Alemtuzumab is FDA-approved for the treatment of some patients with B-cell chronic lymphocytic leukemia (CLL). The use of alemtuzumab to treat MDS, aplastic anemia, or T-cell large granular lymphocytic leukemia is investigational.

Up to 29 participants will take part in this study. All participants will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of MDS (Low, Int-1 by IPSS, or hypocellular) who are either previously untreated or who have been previously treated are eligible for this trial.
2. Patients with the diagnosis of aplastic anemia who have or have not been previously treated are eligible for inclusion if they are not currently candidates for an allogeneic stem cell transplant.
3. Patients with the diagnosis of T-LGL who have or have not been previously treated are eligible for inclusion.
4. Patients must have been off of cytotoxic, immunosuppressive, or targeted therapy (except hydroxyurea) for at least 2 weeks prior to entering this study, and have recovered from the toxic effects of that therapy to grade 1 or less.
5. Adequate organ function as defined: liver function (bilirubin < or = 2mg/dL, AST and/or ALT < or = 3 x ULN) ; kidney function (creatinine < or = 2.5 x ULN ).
6. ECOG performance status of < or = 3.
7. The effects of alemtuzumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
9. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.
10. Patients should have an indication for therapy for their disease such as transfusion dependence or morbidity associated with their cytopenia(s) such as bleeding, severe fatigue, or frequent/multiple infections (eg. neutropenia).

Exclusion Criteria:

1. Pregnant women are excluded from this study because alemtuzumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with alemtuzumab, breastfeeding should be discontinued if the mother is treated with alemtuzumab. These potential risks may also apply to other agents used in this study.
2. Known HIV infection.
3. Known Hepatitis B or Hepatitis C infection.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Patient with documented hypersensitivity to alemtuzumab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 27, 2010 to November 22, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study closed due to slow accrual and change in drug availability.
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [60 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response - Number of Participants Who Achieved Complete Remission (CR)+Partial Remission (PR) - as Per International Working Group (IWG) Response Criteria
Description: Overall response (OR) defined as complete/partial remission for at least 4 weeks or hematologic improvement for at least 8 weeks. Response Criteria are according to the Modified IWG Response Criteria in Myelodysplasia. IWG 2006 response criteria - CR: bone marrow evaluation shows less than or equal to (<=) 5% blasts; normal maturation of all cells lines (mCR), peripheral blood evaluation shows hemoglobin >= 11 gram per deciliter (g/dL), neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts; PR: Same as CR, except blasts decrease by >=50%, still greater than 5% in bone marrow. Hematologic improvement are measured in participants with pretreatment abnormal values: hemoglobin level less than 110 g/L (11 g/dL) or red blood count (RBC)-transfusion dependence, platelet count <100 x 10^9/L or platelet-transfusion dependence, absolute neutrophil count (ANC) less than 1.0 x 10^9/L.
Time Frame: Up to 6 months following treatment; response assessed every 2 months
Population: One subject's response was indeterminate due to the absence of end of therapy assessments.
Measure: Number; unit: participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 6
participants
  Complete Remission (CR) | 0
  Partial Remission (PR) | 0
  Hematologic Improvement | 1
  Disease Progression | 1
  Stable Disease (SD) | 4

ADVERSE EVENTS:
Time Frame: Adverse event collection for 10 day cycle with treatment expected for 3 months.
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=7)
Bacteremia (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=7)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 1 (1)
Elevated AST (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes